CLINICAL TRIAL: NCT07109362
Title: ERP-Based Research on the Modulation of Remimazolam on Working Memory and Brain Network Mechanisms in Glioma Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RM20250717
Record Dates: First submitted 2025-07-17; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Remimazolam Mild Sedation; Healthy Brain and Glioma Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy brain group (Other)
  Interventions: Drug: mild sedation
- Glioma brain group (Other)
  Interventions: Drug: mild sedation

INTERVENTIONS:
Drug: mild sedation — In this experiment, all subjects were administered remimazolam via a TCI pump until they reached a state of mild sedation, as indicated by a MOAA/S score of 4.

SUMMARY:
Remimazolam is a novel ultra-short-acting benzodiazepine with extensive evidence supporting its safety and efficacy in clinical anesthesia and sedation. Its perioperative use in patients with glioma is becoming increasingly common. Glioma is the most common primary intracranial tumor and is often associated with neurocognitive impairment, with memory being the most frequently affected domain. Working memory, which integrates temporary storage and information processing, serves as a cognitive workspace. Currently, the impact of anesthetics on neurocognitive function during the perioperative period in glioma patients remains underexplored. This study aims to investigate the effects of remimazolam-induced mild sedation on working memory in healthy subjects and patients with supratentorial glioma by combining behavioral and electrophysiological measurements, focusing on the relationship with the P3b event-related potential amplitude. Furthermore, it explores how remimazolam sedation influences brain network functional connectivity during the encoding, maintenance, and retrieval phases of memory in healthy individuals and patients with supratentorial glioma.

ELIGIBILITY:
Inclusion Criteria:

A. Healthy brain group:

* Aged 18-65 years;

  * Native speakers of Chinese;

    * Right-handed; ④ Normal vision or corrected vision; ⑤ Healthy brain patient population scheduled for non-neurosurgical operations and anesthesia B. Glioma brain group
* Aged 18-65 years old;

  * Native speakers of Chinese;

    * Right-handed; ④ ASA physical status I-II;

      * Normal vision or corrected vision;

        * Patients with supratentorial glioma who have primary unilateral space-occupying lesions confirmed by CT/MRI and require surgery and anesthesia.

Exclusion Criteria:

A. Healthy brain group:

* Allergic to remimazolam or with contraindications to remimazolam (myasthenia gravis, schizophrenia, severe depressive state);

  * History of drug abuse or alcoholism;

    * History of mental or neurological diseases that prevent cooperation in completing the trial; ④ Pregnant or lactating women;

      * Score of mini-mental state examination (MMSE) < 27; ⑥ Past history of intracranial diseases or intracranial surgery

B. Glioma brain group:

* Receiving sedative treatment within 72 hours prior to the study;

  * Destruction of cerebral structural integrity such as open head injury or cerebral parenchyma resection;

    * Preoperative elevated intracranial pressure requiring mannitol or other intracranial pressure-lowering treatments, or preoperative radiotherapy and chemotherapy;

      * History of drug abuse or alcoholism;

        * Pregnant or lactating women; ⑥ Mini-Mental State Examination (MMSE) score < 27; ⑦ History of allergic reaction to remimazolam or having contraindications to remimazolam. Remimazolam is a national controlled drug with addictive properties and must be used under the guidance of a doctor; ⑧ Those with other mental or neurological diseases who are unable to cooperate in completing the trial; ⑨ Unsuitable for participating in this study due to other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
behavioral results, including reaction time and accuracy rate | All participants completed the working memory test one day before the surgery.
  Participants completed the Sternberg working memory paradigm, with a total of 360 trials. They were required to make yes/no judgments on the memory content, and finally, the accuracy rate and average reaction time will be calculated.
P3b event-related potential (ERP) | All participants completed the working memory test one day before the surgery, with simultaneous collection of 64-channel scalp electroencephalogram (EEG).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided